CLINICAL TRIAL: NCT04273113
Title: Does Heart Rate Variance (HRV) Biofeedback Help Regulate Emotions and Improve Mindfulness in Mentally Unwell Offenders?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-105
Record Dates: First submitted 2020-01-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-09

CONDITIONS: Emotional Dysfunction
Keywords: Biofeedback training, Offenders, Anxiety, Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Rate Variance (HRV) biofeedback training (Experimental): Patients to participate in 15 biofeedback sessions, 3 times a week (5 weeks in total).
  Interventions: Other: Difficulties in Emotional Regulation Scale, Five Facet Mindfulness Questionnaire, Becks Depression and Becks Anxiety; Behavioral: HRV Biofeedback (Healing Rhythms)

INTERVENTIONS:
Other: Difficulties in Emotional Regulation Scale, Five Facet Mindfulness Questionnaire, Becks Depression and Becks Anxiety — Patients asked to complete these 4 questionnaires pre, during and post biofeedback training
Behavioral: HRV Biofeedback (Healing Rhythms) — Sensors placed on fingers to capture heart rate and skin temperature

SUMMARY:
14 participants residing in a forensic psychiatric hospital completed 15 Heart Rate Variance (HRV) biofeedback sessions. They completed 4 psychometric questionnaires, pre, during and post biofeedback training.

DETAILED DESCRIPTION:
This study aimed to establish whether Heart Rate Variance (HRV) biofeedback improved HRV coherence as well as psychological well-being (depression, anxiety, emotion regulation, and mindfulness) over the course of 15 biofeedback sessions in a sample of 14 patients with varying diagnoses; Paranoid Schizophrenia, Schizoaffective Disorder, Personality Disorder or Mixed Diagnosis. All 14 participants (n=10 male, n=4 female) participated in 15 biofeedback sessions. The study was researched and treatment was facilitated by a trainee forensic psychologist working with both male and female offenders residing within a Forensic Psychiatric Hospital, on both low and medium secure wards. An average coherence percentage was captured using the Wild Devine Programme® Relaxing Rhythms software for each session. Quantitative data were collected and analysed before, during and after biofeedback treatment to assess whether there was improvement in psychometric measures of depression, anxiety, emotion regulation and facets of mindfulness. A quasi experimental 'A-B-A design' was employed to assess the research questions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female offenders aged 18 and above.
* Male and female offenders who reside in a medium and low Forensic Psychiatric Hospital.
* Individuals who have the capacity to consent to take part in the research
* Individuals deemed mentally stable and were found to have capacity to consent by their Multi-Disciplinary Team (MDT).

Exclusion Criteria:

* Individuals under the age of 18.
* Individuals who are not detained in a Forensic Psychiatric Hospital.
* Individuals deemed not well enough to consent by their Multi-Disciplinary Team (MDT).
* A level of cognitive impairment determined by diagnosis that would prevent individuals from understanding the feedback obtained. via pictorial or verbal prompts
* Individuals with specific breathing difficulties (e.g., chronic obstructive pulmonary disease) that would restrict them from being able to practice the breathing techniques.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2020-03-28 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotional Regulation (DERS) | 30 minutes (pre, during and post biofeedback training)
  a 36 item self-report questionnaire developed to assess adult difficulties in emotional regulation. six specific dimensions which include; difficulties accepting emotional responses (acceptance), controlling impulse behaviours (impulse), emotional awareness (awareness), emotional clarity (clarity), assessing emotion regulation strategies (strategies) and engaging in goal oriented behaviour when emotionally aroused (goals). Internal consistency for Cronbach's alpha was .93 for the total scale and for DERS-A, .85, DERS-I, .89, DERS-A, .86, DERS-C, .80, DERS-S, .88, and DERS-G, .84
Five Facet Mindfulness Questionnaire (FFMQ) | 30 minutes (pre, during and post biofeedback training)
  Consists of 39 items assessing five facets of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Items are rated on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). The FFMQ has been shown to have good internal consistency and significant relationships in the predicted directions with a variety of constructs related to mindfulness. The internal consistencies (Cronbach α) for these facets have been reported as 0.75 for FFMQ-NR, 0.83 for FFMQ-O, 0.87 for FFMQ-A, 0.91 for FFMQ-D, and 0.87 for FFMQ-NJ
Becks Depression Inventory (BDI-II) | 15 minutes (pre, during and post biofeedback training)
  A 21-item self-report scale that surveys common symptoms of depression on a 4-point scale ranging from 0 to 3. Internal consistency of the BDI-II was demonstrated to be good (Cronbach's α=.91; Beck, Steer, Ball et al., 1996) and the 1-week test-retest reliability was shown to be high.
Becks Anxiety Inventory (BAI) | 15 minutes (pre, during and post biofeedback training)
  Consists of 21 statements used to measure the severity of an individual's anxiety. When completing the BAI, individuals rate the severity of each symptom on a 4-point scale ranging from 0 (not at all) to 3 (severely-I could barely stand it). Good internal consistency (Cronbach's α=.92) and test-retest reliability (r=.75).

SECONDARY OUTCOMES:
Heart Rate Variance (HRV) biofeedback | 10 minutes per session
  Heart rate coherence scores were assessed using the IoM butterfly Grapher. The coherence score is based upon a composite score of 0-100%; 0 being no coherence, 100% being perfect coherence.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina V Atkinson, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No